CLINICAL TRIAL: NCT00706589
Title: A Randomized, Double-blind, Dose-adjustment, Placebo-controlled Study to Evaluate the Efficacy and Safety of Aripiprazole in Children and Adolescents With Chronic Tic Disorders or Tourette's Disorder
Brief Title: Aripiprazole in Children and Adolescents With Chronic Tic Disorder or Tourette's Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 031-KOA-0703
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2013-07-26 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Motor or Vocal Tic Disorder; Tourette's Disorder
Keywords: Chronic Motor Tic disorder; Chronic Phonic Tic disorder; Tourette's disorder; Aripiprazole; Abilify; Children; Adolescent
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Aripiprazole 2mg,5mg,10mg,15mg,20mg orally administrated Once a day (Titration according to the protocol)
  Interventions: Drug: aripiprazole
- 2 (Placebo Comparator): Placebo 2mg,5mg,10mg,15mg,20mg orally administrated Once a day (Titration according to the protocol)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: aripiprazole — Initial dose : 2mg, Maximum dose : 20mg
  Other Names: Abilify
  Arms: 1
Drug: placebo — Initial dose: 2mg, Maximum dose:20mg
  Arms: 2

SUMMARY:
The purpose of this trial is to demonstrate the efficacy and safety of aripiprazole in children and adolescents aged 6~18 years with chronic tic disorders or Tourette's disorder

ELIGIBILITY:
Inclusion Criteria:

1. Patients who can provide an assent form signed by themselves and informed consent form by their legal representatives prior to performing of any study procedures.
2. Male or female children and adolescents aged 6 to 18 years
3. Patients who are diagnosed with chronic tic disorders(Motor or Phonic) or Tourette's disorder according to DSM-IV(Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition)(using K-SADS-PL-K (Kiddle-Schedule for Affective Disorders and Schizophrenia,Present and Lifetime Version-Korean version)) and require drug therapy.
4. The total tic score of the K-YGTSS (Korean version of Yale Global Tic Severity Scale)is more than 22 at baseline

Exclusion Criteria:

1. Patients with secondary tic symptoms accompanied by Tardive tics, Huntington disease, neuroacanthocytosis, mental retardation, or autism
2. Patients with IQ (Intelligence quotient) (assessed using KEDI-WISC (Korean educational Development Institute-Wechsler Intelligence Scale for children)) 70 and lower than 70
3. Patients with a history of neuroleptic malignant syndrome
4. Patients with antipsychotic or alcohol use disorder (abuse, dependence, and/or withdrawal) according to DSM-IV criteria for the past 3 months
5. Patients with a history of allergy or hypersensitivity reaction to aripiprazole
6. Patients with a history of resistance to treatment with antipsychotics
7. Patients who have participated in another clinical study within 1 month prior to screening
8. Patients who have previously taken aripiprazole or participated in a clinical study with aripiprazole

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soochurl Cho, MD. Ph.D, Principal Investigator — Seoul National University Hospital
Locations (6):
- South Korea (6):
  - Inha University Hospital, Inchon
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Chung-Ang Univ. Medical center, Seoul

REFERENCES:
- [Derived] Yoo HK, Joung YS, Lee JS, Song DH, Lee YS, Kim JW, Kim BN, Cho SC. A multicenter, randomized, double-blind, placebo-controlled study of aripiprazole in children and adolescents with Tourette's disorder. J Clin Psychiatry. 2013 Aug;74(8):e772-80. doi: 10.4088/JCP.12m08189. PMID 24021518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period :Aug2008~Jan2010 Types of location: Medical Center
Pre-assignment Details: antipsychotic or antiparkinson drugs should be washed out 1~2 weeks prior to randomization.
Groups:
- Aripiprazole: Aripiprazole 2mg,5mg,10mg,15mg, 20mg orally administrated Once a day (Titration according to the protocol) Mode of administration: P.O
- Placebo: Placebo 2mg,5mg,10mg,15mg, 20mg orally administrated Once a day (Titration according to the protocol)10mg,15mg, 20mg Mode of administration: P.O
Period: Overall Study
Arm/Group | Aripiprazole | Placebo
Started | 32 | 29
Completed | 29 | 25
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Aripiprazole: Aripiprazole 2mg,5mg,10mg,15mg
- Placebo: Placebo 2mg,5mg,10mg,15mg
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 29 | 61
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 10.97 (2.49) | 10.93 (3.00) | 10.95 (2.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 30 | 23 | 53
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 32 | 29 | 61

OUTCOME MEASURES:

1. Secondary Outcome: 1)Percent Change of Total Tic Scores on the Korean Version of YaleGlobalTicseverity Scale.2)Response Rate Assessed With the Tic Score ClinicalGlobalImpressionImprovementScale.3)Mean Change in Scores on the Tic Score ClinicalGlobal ImpressionSeverityScale.
Time Frame: 10 weeks
Reporting Status: Not Posted
Measure: Mean; unit: participants

2. Primary Outcome: Mean Change of Total Tic Scores in K-YGTSS From Randomization (Baseline, Visit 2) to the Final Visit (Visit 7)
Description: The meaning of the total tic scores is a sum of the total motor tic score and total phonic tic score and the total tic score will be indicated from zero point to 50 points. And also, for the global tic severity scale is sum of the total tic scores and impairment score and it will be indicated from zero point to 100 points. Additionally, for the imparment score is also indicated from zero to 50 points same as total tic scores. And it is divided as 0 point, 10 point, 20 point and etc… Lastly, someone who gets a high score, it will be considered worse result.
Time Frame: 10 week
Population: ITT (Intention-To-Treat)analysis
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Aripiprazole: Aripiprazole 2mg,5mg,10mg,15mg, 20mg
- Placebo: Placebo 2mg,5mg,10mg,15mg, 20mg
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 31 | 29
units on a scale | -9.62 [-32 to 8] | -14.97 [-33 to 2]

ADVERSE EVENTS:
Time Frame: 14 week
Description: A total of 60 subjects were included in the safety analysis; 28 in Placebo group and 32 in Aripiprazole group. Note that one subject who was randomized to Placebo group but took Aripiprazole due to prescription error was included in Aripiprazole group as per the actual administration for the safety analysis.
Arm/Group | Aripiprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/28
Other Adverse Events (participants affected / at risk) | 24/32 | 20/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=32) | Placebo (N=28)
Sedation (Nervous system disorders) | 4 (5) | 3 (5)
Akathisia (Nervous system disorders) | 2 (2) | 4 (5)
Headache (Nervous system disorders) | 5 (5) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4)
Extrapyramidal disorder (Nervous system disorders) | 3 (3) | 2 (2)
Somnolence (Nervous system disorders) | 4 (5) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4)
Nasopharyngitis (Infections and infestations) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (4)
Irritability (General disorders) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other